CLINICAL TRIAL: NCT03367104
Title: Electrical Dyssynchrony in Narrow QRS Heart Failure Patients as Assessed by the ECG Belt
Brief Title: Narrow QRS HF Patients Assessed by ECG Belt
Status: Completed | Type: Observational
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Alan J. Bank, MD, Medical Director of Research - UHVC, Allina Health System
Other Study IDs: ERP 3771
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Normal healthy controls
  Interventions: Device: ECG Belt
- Heart failure patients
  Interventions: Device: ECG Belt

INTERVENTIONS:
Device: ECG Belt — Assess electrical dyssynchrony with an anterior-posterior body surface mapping system.

SUMMARY:
The purpose of this study is to quantitate electrical dyssynchrony in heart failure (HF) patients with a narrow QRS complexes (≤ 130 ms) using the ECG Belt. This is a pilot study that is designed to provide data that can be used in designing and implementing a prospective study of cardiac resynchronization therapy (CRT) in narrow QRS patients selected and optimized using the ECG Belt.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or their legal guardian) must be willing to provide informed consent for their participation in the study
* Subject ≥ 18 years old

Exclusion Criteria:

* Subject has unhealed-open wounds on the torso and/or has a history of severe allergic reactions from ECG electrode gel
* Subject is enrolled in a concurrent study that could confound the results of this study
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and those with heart failure (reduced ejection fraction) with QRS duration ≤ 130 ms.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Electrical dyssynchrony quantification | through acute study completion (~60 minutes)
  Collect ECG data with ECG Belt

CONTACTS AND LOCATIONS:
Overall Officials: Alan Bank, MD, Principal Investigator — Allina Health System
Locations (1):
- United Heart & Vascular Clinic, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No